CLINICAL TRIAL: NCT01259128
Title: A Phase III Randomized, Open-Label, Multicenter Study to Investigate the Safety and Pharmacokinetics of SER120 Nasal Spray Formulations in Elderly Patients (≥ 75 Years Old) With Nocturia
Brief Title: Study to Investigate the Safety and Pharmacokinetics of SER120 Nasal Spray in Elderly Patients With Nocturia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Serenity Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SPC-SER120-ELD-2010-01
Record Dates: First submitted 2010-04-22; First posted 2010-12-13 (Estimated); Results first posted 2020-11-17 (Actual); Last update posted 2020-11-17 (Actual); Status verified 2014-04

CONDITIONS: Nocturia
MeSH Terms: conditions — Nocturia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- SER120 500 ng/day (Experimental): SER120 Level 1 (500 ng/day)
  Interventions: Drug: SER120 Nasal Spray 500 ng/day
- SER120 750 ng/day (Experimental): SER120 Level 2 (750 ng/day)
  Interventions: Drug: SER120 nasal spray 750 ng/day

INTERVENTIONS:
Drug: SER120 Nasal Spray 500 ng/day — SER120 Level 1
  Arms: SER120 500 ng/day
Drug: SER120 nasal spray 750 ng/day — SER120 (750 ng/day)
  Arms: SER120 750 ng/day

SUMMARY:
The purpose of this study is to determine if SER120 nasal spray is well tolerated in 75 years or older nocturic patients.

DETAILED DESCRIPTION:
Patients entering the study are randomized to either Level 1 SER120 nasal spray concentration or Level 2 SER120 nasal spray concentration

ELIGIBILITY:
Inclusion Criteria:

* Male & female greater or equal to 75 years of age, history of nocturia

Exclusion Criteria:

* CHF, Diabetes, Diabetes Insipidus, Renal Insufficiency, Heptatic Insufficiency, Incontinence, Illness requiring steroid, current or past urologic maliganancy, nephrotic syndrome
* Unexplained pelvic masses
* Urinary bladder surgery or radiotherapy
* Sleep apnea

Ages: 75 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 32 (Actual)
Dates: Start 2010-04; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Dr. Jolene Berg, San Antonio, Texas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- SER120 500 ng: All participants received 500 ng once daily
- SER120 750 ng: All participants received 750 ng once daily
Period: Overall Study
Arm/Group | SER120 500 ng | SER120 750 ng
Started | 15 | 17
Completed | 15 | 15
Not Completed | 0 | 2

BASELINE CHARACTERISTICS:
Population: ITT
Groups:
- Total: Total of all reporting groups
Arm/Group | SER120 500 ng | SER120 750 ng | Total
Number analyzed (Participants) | 15 | 16 | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 79 (3.6) | 79.1 (3.3) | 79.1 (3.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 10 | 11 | 21
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 14 | 16 | 30
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15 | 16 | 31

OUTCOME MEASURES:

1. Primary Outcome: Serum Sodium Levels at Baseline and During Treatment
Description: Mean serum sodium reported at baseline, Day 4, Day 8, Day 15, Day 22, Day 29, Day 43 and Day 57.
Time Frame: baseline, Day 4, Day 8, Day 15, Day 22, Day 29, Day 43 and Day 57
Population: Safety population
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | SER120 500 ng | SER120 750 ng
Number analyzed (Participants) | 15 | 17
mmol/L
  Baseline | 141.0 (2.4) | 140.0 (1.7)
  Day 4 | 139.2 (3.0) | 140.3 (1.3)
  Day 8 | 139.1 (3.2) | 140.4 (1.8)
  Day 15 | 140.4 (2.1) | 140.2 (1.4)
  Day 22 | 139.5 (3.2) | 140.0 (1.4)
  Day 29 | 139.7 (2.7) | 139.7 (2.1)
  Day 43 | 139.9 (2.7) | 139.6 (1.5)
  Day 57 | 140.9 (2.6) | 141.1 (1.7)

2. Secondary Outcome: Change in Mean Nocturic Episodes Per Night
Description: Change in mean nocturic episodes per night between baseline and Week 8
Time Frame: Mean value at Week 8 minus mean value at baseline
Population: Intent-to-Treat Population
Measure: Mean (Standard Deviation); unit: nocturic episodes per night
Arm/Group | SER120 500 ng | SER120 750 ng
Number analyzed (Participants) | 15 | 16
nocturic episodes per night | -1.5 (0.8) | -1.4 (0.7)

3. Secondary Outcome: Percent of Participants With Greater or Equal to 50% Reduction in the Number of Nocturic Episodes
Description: Percent of participants with greater or equal to 50% reduction in number of nocturic episodes at Week 8 compared to Baseline
Time Frame: 8 weeks
Population: Intent-To-Treat Polpulation
Measure: Count of Participants; unit: Participants
Arm/Group | SER120 500 ng | SER120 750 ng
Number analyzed (Participants) | 15 | 16
Participants | 11 | 11

ADVERSE EVENTS:
Time Frame: 8 Weeks
Description: Safety Population
Arm/Group | SER120 500 ng | SER120 750 ng
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/17
Other Adverse Events (participants affected / at risk) | 8/15 | 12/17
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SER120 500 ng (N=15) | SER120 750 ng (N=17)
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
lacrimation increased (Eye disorders) | 1 (1) | 2 (2)
abnormal sensation in eye (Eye disorders) | 1 (1) | 0 (0)
diarrhea (Gastrointestinal disorders) | 2 (2) | 0 (0)
abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
chapped lips (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0)
gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
gingival pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
hypoaesthesia oral (Gastrointestinal disorders) | 1 (1) | 0 (0)
oral pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Chills (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (1)
sensation of pressure (General disorders) | 1 (1) | 0 (0)
nasopharyngitis (Infections and infestations) | 1 (1) | 1 (1)
Excoriation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Incisional hernia (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Joint sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
headache (Nervous system disorders) | 1 (1) | 1 (1)
dizziness (Nervous system disorders) | 1 (1) | 0 (0)
urinary hesitation (Renal and urinary disorders) | 0 (0) | 1 (1)
nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 6 (6)
sneezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4)
rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
rhinalgia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
paranasal sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
sinus disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
sebaceous cyst excision (Surgical and medical procedures) | 0 (0) | 1 (1)
skin cosmetic procedure (Surgical and medical procedures) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes